CLINICAL TRIAL: NCT00784615
Title: Descriptive, Transversal Study of Evaluation of Cardiovascular Risks Factors and Prevalence of Metabolic Syndrome in the Different Phenotypes of Women With Polycystic Ovary Syndrome
Brief Title: Evaluation of Endocrine and Metabolic Parameters in the New Diagnostic Phenotypes of Polycystic Ovary Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidad Nacional de Córdoba (Other)
Collaborators: Fundación Florencio Fiorini (Unknown)
Responsible Party: Carolina Fux Otta, Hospital Universitario de Maternidad y Neonatología. UNC
Other Study IDs: Fux-2
Record Dates: First submitted 2008-11-03; First posted 2008-11-04 (Estimated); Last update posted 2008-11-19 (Estimated); Status verified 2008-10

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Phenotypes of Polycystic Ovary Syndrome; Cardiovascular risk factors; Adiponectin; C Reactive Protein
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- 1: Women with polycystic ovaries, oligo or anovulation and hyperandrogenism.
  Interventions: Procedure: Blood samples, transvaginal ultrasound
- 2: Women with polycystic ovaries and oligo or anovulation without hyperandrogenism
  Interventions: Procedure: Blood samples, transvaginal ultrasound
- 3: Women with normal ovaries, oligo or anovulation and hyperandrogenism
  Interventions: Procedure: Blood samples, transvaginal ultrasound
- 4: Women with normal ovaries, oligo or anovulation and hyperandrogenism
  Interventions: Procedure: Blood samples, transvaginal ultrasound
- 5: Women with out polycystic ovary syndrome
  Interventions: Procedure: Blood samples, transvaginal ultrasound

INTERVENTIONS:
Procedure: Blood samples, transvaginal ultrasound — Total testosterone, bioavailable testosterone, Free androgen index, Total cholesterol, LDL Cholesterol, HDL Cholesterol, Triglycerides, insulinemia, OGTT, HOMA index, Adiponectin, C Reactive Protein

SUMMARY:
Polycystic ovary syndrome (PCOS) is a very frequent endocrine disease of women in reproductive age, with an estimated prevalence of 5 to 10 % according to the studied population. In 2003 a committee of experts joined in Rotterdam under the auspice of the American Society for Reproductive Medicine and the European Society for Human Reproduction and Embryology, defined diagnostic criteria. It should include unless two of the following: menstrual irregularities; excess of male hormones (clinic or biochemical) and polycystic ovaries under ultrasound examination; giving rise to four subgroups or phenotypes:

1- Women with polycystic ovaries, hyperandrogenism and oligoamenorrhea . 2. Women with normal ovaries, hyperandrogenism and oligoamenorrhea. 3- Women with polycystic ovaries, oligoamenorrhea without hyperandrogenism. 4- Women with polycystic ovaries, hyperandrogenism with normal menses. PCOS shares components of Metabolic Syndrome for the high prevalence of insulin resistance (abdominal obesity, impaired glucose tolerance, type 2 diabetes, hypertension, endothelial dysfunction, impaired lipid profile and probably cardiovascular disease). All these findings lead us to assume that women with PCOS could have an increased risk of developing cardiovascular disease. Nevertheless it is premature to assume that every PCOS phenotype has the same cardiac and metabolic risk factors. So, it is important to evaluate the endocrine and metabolic characteristic in different phenotypes of PCOS to prevent the co morbidities that predispose to cardiovascular disease. And of course to avoid unnecessary measures in groups that could not show increased risk.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is a very frequent endocrine disease of women in reproductive age, with an estimated prevalence of 5 to 10 % according to the studied population.

Its cause remains not fully understood. PCOS is characterized by hyperandrogenism, chronic anovulation and / or polycystic ovaries. Patients, in a high percentage of cases show obesity, hirsutism, acne, menstrual irregularities and infertility. Clinically and biologically PCOS is a heterogeneous disorder with a not yet clear pathogenesis. Therefore, discussions on its definition and diagnosis still subsist. Seventy years ago Stein and Leventhal published their findings in 7 women with amenorrhea, hirsutism, acne, obesity and polycystic appearance of their ovaries. Since then, diagnostic criteria for PCOS suffered multiple modifications.

In 1990 a group of experts under the auspices of the National Institutes of Health (NIH) considered affected by PCOS every woman with hyperandrogenism and chronic anovulation; after having excluded other specific diseases that mimic that clinic like Cushing's syndrome, androgen secreting tumors and congenital adrenal hyperplasia (NIH criteria). The presence of polycystic ovaries under ultrasound exploration was considered controversial criteria and was not included for diagnosis. In May 2003 a new committee of experts joined in Rotterdam under the auspice of the American Society for Reproductive Medicine (ASRM) and the European Society for Human Reproduction and Embryology (ESHRE), included polycystic ovaries by ultrasound to the physiologic abnormalities for diagnosis. Thus, diagnosis should include unless two of the following: oligo or anovulation; hyperandrogenism (clinic or biochemical) and polycystic ovaries under ultrasound examination.

Rotterdam consensus widened the definition already proposed by NIH in 1990 giving rise to four subgroups or phenotypes:

1- Women with polycystic ovaries, hyperandrogenism and oligoamenorrhea. 2. Women with normal ovaries, hyperandrogenism and oligoamenorrhea. 3- Women with polycystic ovaries, oligoamenorrhea without hyperandrogenism. 4- Women with polycystic ovaries, hyperandrogenism with normal menses. This new criteria increase de prevalence, diversity and also controversy about PCOS. Some authors like Franks accept that the new consensus gave significant advances in the etiological knowledge of the syndrome. Others, like Azziz, proposed that is premature to include ovulating women and the ones with no clear evidence of androgens excess. In the last subgroups is no clear if they have an increased risk of cardiovascular and / or metabolic diseases.

The clinical heterogeneity of the syndrome is the product of a multifaceted process; where converge genetic and environmental influences. Many hypotheses try to explain the primary defect; but insulin resistance (IR) seems the most suitable according to most of studies. IR is present in 60 to 70 % of patients independently of obesity. Compensatory hyperinsulinism has a fundamental role in the pathology of PCOS. In vitro insulin stimulates androgen synthesis in ovary theca cells, acting on its own receptor and inhibits hepatic synthesis of sex hormone binding globulin (SHBG), increasing free testosterone. It also leads to the amplification of LH induced expression of cytochrome P450c 17 alfa (a limiting enzyme in androgen synthesis).

PCOS shares components of Metabolic Syndrome for the high prevalence of IR (abdominal obesity, impaired glucose tolerance, type 2 diabetes, hypertension, endothelial dysfunction, impaired lipid profile and probably cardiovascular disease). Dunaif and Sam using NIH criteria for PCOS diagnosis suggested a sole entity called XX syndrome. Central adiposity seems to play an important role in the development of this metabolic phenotype trough the production of many cytokines and adipocytes derived proteins, known as "adipocytokines". Failures on its regulation could contribute to the development of IR. The late one for itself or trough metabolic disturbances is associated with endothelial dysfunction and atherosclerosis.

Adiponectin is exclusively secreted in adipose tissue and could inhibit the expression of vascular endothelial adhesion molecules induced by TNF-alfa. So, it could be an anti atherogenic effect of adiponectin. In obese subjects and those with type 2 diabetes and IR (whom has a high incidence of coronary atherosclerosis) it was found low plasma levels of adiponectin. Recent studies propose low serum levels of adiponectin as an early marker for metabolic risk in women with PCOS.

C Reactive Protein (CRP), a low grade inflammation marker, has been suggested as an independent predictor of cardiovascular event in women; even more relevant than LDL cholesterol. Those facts have been reassured in the recent publication of Reynolds risk score which adds to the classical ATP III´s Framingham score; the usage of CRP in women, increasing its prognostic value. Higher levels of CRP have been described in women with PCOS compared with normal controls.

All these findings lead us to assume that women with PCOS have an increased risk of developing cardiovascular disease. As there is no universally accepted definition for PCOS, studies that show an association between PCOS and cardiovascular disease are of relative value. Legro stated that "It is premature to assume that every PCOS phenotype has the same cardiac and metabolic risk factors".

So, it is important to evaluate the endocrine and metabolic characteristic in different phenotypes of PCOS to prevent the co morbidities that predispose to cardiovascular disease. And of course to avoid unnecessary measures in groups that could not show increased risk.

ELIGIBILITY:
Inclusion Criteria:

Two of the following

* Ovulatory Dysfunction: Clinically defined by oligomenorrhea (menstrual cycles lasting more than 35 days) or amenorrhea (lacking of menstruations in the last 90 days). In patients with menstrual cycles between 25 and 35 days, a serum level of progesterone drawn during days 21 to 23 of cycle < a 4 ng/ml.
* Clinical hyperandrogenism defined for the presence of hirsutism, acne, androgenic alopecia) and or biochemical (increases in total testosterone, bioavailable testosterone or free androgen index).
* Polycystic Ovaries: Defined by the presence, in as less one ovary, of 12 or more follicles (measuring 2 to 9 mm in diameter) and or increased ovarian volume > 10 mL).

Exclusion Criteria:

* Hyperprolactinemia
* Hypothyroidism
* Other causes of hyperandrogenism like Cushing's Syndrome, congenital adrenal hyperplasia, androgens secreting tumors
* Drug therapy used three months previous to enrollment in the study

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women in reproductive age with diagnosis of polycystic ovary syndrome according to Rotterdam criteria
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2007-12

PRIMARY OUTCOMES:
Serum levels: Total, bioavailable testosterone, Free androgen index. Total, LDL and HDL Cholesterol, Triglycerides, insulinemia, OGTT, HOMA index, Adiponectin, C Reactive Protein. Transvaginal Ultrasound:Number,size of ovary follicles and ovary volume | At the begining of the study

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Fux Otta, MD, Principal Investigator — Hospital Universitario de Maternidad y Neonatología. Universidad Nacional de Córdoba; Marta Fiol de Cuneo, MD, Study Director — Catedra de Fisiología Humana. Universidad Nacional de Córdoba
Locations (1):
- Hospital Universitario de Maternidad y Neonatología, Córdoba, Córdoba Province, Argentina

REFERENCES:
- [Background] Alberti KG, Zimmet P, Shaw J; IDF Epidemiology Task Force Consensus Group. The metabolic syndrome--a new worldwide definition. Lancet. 2005 Sep 24-30;366(9491):1059-62. doi: 10.1016/S0140-6736(05)67402-8. No abstract available. PMID 16182882
- [Background] Asuncion M, Calvo RM, San Millan JL, Sancho J, Avila S, Escobar-Morreale HF. A prospective study of the prevalence of the polycystic ovary syndrome in unselected Caucasian women from Spain. J Clin Endocrinol Metab. 2000 Jul;85(7):2434-8. doi: 10.1210/jcem.85.7.6682. PMID 10902790
- [Background] Azziz R, Woods KS, Reyna R, Key TJ, Knochenhauer ES, Yildiz BO. The prevalence and features of the polycystic ovary syndrome in an unselected population. J Clin Endocrinol Metab. 2004 Jun;89(6):2745-9. doi: 10.1210/jc.2003-032046. PMID 15181052
- [Background] Azziz R. Controversy in clinical endocrinology: diagnosis of polycystic ovarian syndrome: the Rotterdam criteria are premature. J Clin Endocrinol Metab. 2006 Mar;91(3):781-5. doi: 10.1210/jc.2005-2153. Epub 2006 Jan 17. PMID 16418211
- [Background] Barbieri RL, Makris A, Randall RW, Daniels G, Kistner RW, Ryan KJ. Insulin stimulates androgen accumulation in incubations of ovarian stroma obtained from women with hyperandrogenism. J Clin Endocrinol Metab. 1986 May;62(5):904-10. doi: 10.1210/jcem-62-5-904. PMID 3514651
- [Background] Bloomgarden ZT. American Association of Clinical Endocrinologists (AACE) consensus conference on the insulin resistance syndrome: 25-26 August 2002, Washington, DC. Diabetes Care. 2003 Apr;26(4):1297-303. doi: 10.2337/diacare.26.4.1297. No abstract available. PMID 12663612
- [Background] Boulman N, Levy Y, Leiba R, Shachar S, Linn R, Zinder O, Blumenfeld Z. Increased C-reactive protein levels in the polycystic ovary syndrome: a marker of cardiovascular disease. J Clin Endocrinol Metab. 2004 May;89(5):2160-5. doi: 10.1210/jc.2003-031096. PMID 15126536
- [Background] Christian RC, Dumesic DA, Behrenbeck T, Oberg AL, Sheedy PF 2nd, Fitzpatrick LA. Prevalence and predictors of coronary artery calcification in women with polycystic ovary syndrome. J Clin Endocrinol Metab. 2003 Jun;88(6):2562-8. doi: 10.1210/jc.2003-030334. PMID 12788855
- [Background] Dahlgren E, Janson PO, Johansson S, Lapidus L, Oden A. Polycystic ovary syndrome and risk for myocardial infarction. Evaluated from a risk factor model based on a prospective population study of women. Acta Obstet Gynecol Scand. 1992 Dec;71(8):599-604. doi: 10.3109/00016349209006227. PMID 1336918
- [Background] Diamanti-Kandarakis E, Kouli CR, Bergiele AT, Filandra FA, Tsianateli TC, Spina GG, Zapanti ED, Bartzis MI. A survey of the polycystic ovary syndrome in the Greek island of Lesbos: hormonal and metabolic profile. J Clin Endocrinol Metab. 1999 Nov;84(11):4006-11. doi: 10.1210/jcem.84.11.6148. PMID 10566641
- [Background] Dunaif A. Insulin resistance and the polycystic ovary syndrome: mechanism and implications for pathogenesis. Endocr Rev. 1997 Dec;18(6):774-800. doi: 10.1210/edrv.18.6.0318. PMID 9408743
- [Background] Dunaif A, Segal KR, Futterweit W, Dobrjansky A. Profound peripheral insulin resistance, independent of obesity, in polycystic ovary syndrome. Diabetes. 1989 Sep;38(9):1165-74. doi: 10.2337/diab.38.9.1165. PMID 2670645
- [Background] Ehrmann DA. Polycystic ovary syndrome. N Engl J Med. 2005 Mar 24;352(12):1223-36. doi: 10.1056/NEJMra041536. No abstract available. PMID 15788499
- [Background] Ehrmann DA, Barnes RB, Rosenfield RL, Cavaghan MK, Imperial J. Prevalence of impaired glucose tolerance and diabetes in women with polycystic ovary syndrome. Diabetes Care. 1999 Jan;22(1):141-6. doi: 10.2337/diacare.22.1.141. PMID 10333916
- [Background] Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults. Executive Summary of The Third Report of The National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, And Treatment of High Blood Cholesterol In Adults (Adult Treatment Panel III). JAMA. 2001 May 16;285(19):2486-97. doi: 10.1001/jama.285.19.2486. No abstract available. PMID 11368702
- [Background] FERRIMAN D, GALLWEY JD. Clinical assessment of body hair growth in women. J Clin Endocrinol Metab. 1961 Nov;21:1440-7. doi: 10.1210/jcem-21-11-1440. No abstract available. PMID 13892577
- [Background] Franks S. Controversy in clinical endocrinology: diagnosis of polycystic ovarian syndrome: in defense of the Rotterdam criteria. J Clin Endocrinol Metab. 2006 Mar;91(3):786-9. doi: 10.1210/jc.2005-2501. Epub 2006 Jan 17. PMID 16418209
- [Background] Franks S, Gharani N, Waterworth D, Batty S, White D, Williamson R, McCarthy M. The genetic basis of polycystic ovary syndrome. Hum Reprod. 1997 Dec;12(12):2641-8. doi: 10.1093/humrep/12.12.2641. PMID 9455828
- [Background] Kelly CC, Lyall H, Petrie JR, Gould GW, Connell JM, Sattar N. Low grade chronic inflammation in women with polycystic ovarian syndrome. J Clin Endocrinol Metab. 2001 Jun;86(6):2453-5. doi: 10.1210/jcem.86.6.7580. PMID 11397838
- [Background] Kershaw EE, Flier JS. Adipose tissue as an endocrine organ. J Clin Endocrinol Metab. 2004 Jun;89(6):2548-56. doi: 10.1210/jc.2004-0395. PMID 15181022
- [Background] Legro RS. The genetics of polycystic ovary syndrome. Am J Med. 1995 Jan 16;98(1A):9S-16S. doi: 10.1016/s0002-9343(99)80053-9. PMID 7825646
- [Background] Legro RS. Polycystic ovary syndrome and cardiovascular disease: a premature association? Endocr Rev. 2003 Jun;24(3):302-12. doi: 10.1210/er.2003-0004. PMID 12788801
- [Background] Legro RS, Kunselman AR, Dunaif A. Prevalence and predictors of dyslipidemia in women with polycystic ovary syndrome. Am J Med. 2001 Dec 1;111(8):607-13. doi: 10.1016/s0002-9343(01)00948-2. PMID 11755503
- [Background] Ludwig E. Androgenetic alopecia. Arch Dermatol. 1977 Jan;113(1):109. doi: 10.1001/archderm.1977.01640010111023. No abstract available. PMID 831614
- [Background] Nestler JE, Powers LP, Matt DW, Steingold KA, Plymate SR, Rittmaster RS, Clore JN, Blackard WG. A direct effect of hyperinsulinemia on serum sex hormone-binding globulin levels in obese women with the polycystic ovary syndrome. J Clin Endocrinol Metab. 1991 Jan;72(1):83-9. doi: 10.1210/jcem-72-1-83. PMID 1898744
- [Background] Norman RJ, Homan G, Moran L, Noakes M. Lifestyle choices, diet, and insulin sensitizers in polycystic ovary syndrome. Endocrine. 2006 Aug;30(1):35-43. doi: 10.1385/ENDO:30:1:35. PMID 17185790
- [Background] Ouchi N, Kihara S, Arita Y, Maeda K, Kuriyama H, Okamoto Y, Hotta K, Nishida M, Takahashi M, Nakamura T, Yamashita S, Funahashi T, Matsuzawa Y. Novel modulator for endothelial adhesion molecules: adipocyte-derived plasma protein adiponectin. Circulation. 1999 Dec 21-28;100(25):2473-6. doi: 10.1161/01.cir.100.25.2473. PMID 10604883
- [Background] Orio F Jr, Palomba S, Cascella T, Milan G, Mioni R, Pagano C, Zullo F, Colao A, Lombardi G, Vettor R. Adiponectin levels in women with polycystic ovary syndrome. J Clin Endocrinol Metab. 2003 Jun;88(6):2619-23. doi: 10.1210/jc.2002-022033. PMID 12788865
- [Background] Paradisi G, Steinberg HO, Hempfling A, Cronin J, Hook G, Shepard MK, Baron AD. Polycystic ovary syndrome is associated with endothelial dysfunction. Circulation. 2001 Mar 13;103(10):1410-5. doi: 10.1161/01.cir.103.10.1410. PMID 11245645
- [Background] Ridker PM, Buring JE, Cook NR, Rifai N. C-reactive protein, the metabolic syndrome, and risk of incident cardiovascular events: an 8-year follow-up of 14 719 initially healthy American women. Circulation. 2003 Jan 28;107(3):391-7. doi: 10.1161/01.cir.0000055014.62083.05. PMID 12551861
- [Background] Ridker PM, Rifai N, Rose L, Buring JE, Cook NR. Comparison of C-reactive protein and low-density lipoprotein cholesterol levels in the prediction of first cardiovascular events. N Engl J Med. 2002 Nov 14;347(20):1557-65. doi: 10.1056/NEJMoa021993. PMID 12432042
- [Background] Robinson S, Henderson AD, Gelding SV, Kiddy D, Niththyananthan R, Bush A, Richmond W, Johnston DG, Franks S. Dyslipidaemia is associated with insulin resistance in women with polycystic ovaries. Clin Endocrinol (Oxf). 1996 Mar;44(3):277-84. doi: 10.1046/j.1365-2265.1996.674495.x. PMID 8729522
- [Background] Rotterdam ESHRE/ASRM-Sponsored PCOS Consensus Workshop Group. Revised 2003 consensus on diagnostic criteria and long-term health risks related to polycystic ovary syndrome. Fertil Steril. 2004 Jan;81(1):19-25. doi: 10.1016/j.fertnstert.2003.10.004. PMID 14711538
- [Background] Sam S, Dunaif A. Polycystic ovary syndrome: syndrome XX? Trends Endocrinol Metab. 2003 Oct;14(8):365-70. doi: 10.1016/j.tem.2003.08.002. PMID 14516934
- [Background] Talbott E, Clerici A, Berga SL, Kuller L, Guzick D, Detre K, Daniels T, Engberg RA. Adverse lipid and coronary heart disease risk profiles in young women with polycystic ovary syndrome: results of a case-control study. J Clin Epidemiol. 1998 May;51(5):415-22. doi: 10.1016/s0895-4356(98)00010-9. PMID 9619969
- [Background] Wild RA. Long-term health consequences of PCOS. Hum Reprod Update. 2002 May-Jun;8(3):231-41. doi: 10.1093/humupd/8.3.231. PMID 12078834
- [Background] Sir-Petermann T, Maliqueo M, Codner E, Echiburu B, Crisosto N, Perez V, Perez-Bravo F, Cassorla F. Early metabolic derangements in daughters of women with polycystic ovary syndrome. J Clin Endocrinol Metab. 2007 Dec;92(12):4637-42. doi: 10.1210/jc.2007-1036. Epub 2007 Sep 11. PMID 17848407
- See also: Funding non profit organization — http://www.fff.org.ar